CLINICAL TRIAL: NCT05088018
Title: A Placebo-controlled, Triple-blind, Pre-post Interventional Study of Swallowable Cannabigerol Tablets on Sleep Quality in Veterans
Brief Title: Swallowable Cannabigerol Tablets for Sleep Quality In Veterans (Veterans Exploring Cannabigerol for Sleep)
Acronym: ECS21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chris Emerson (Industry)
Collaborators: Veterans Cannabis Group (Unknown); Curebase Inc. (Industry); Santa Cruz Veterans Alliance (Unknown)
Responsible Party: Sponsor-Investigator, Chris Emerson, CEO & Founder, Metta Medical, Inc
Organization: Metta Medical, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VetsECS21
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Sleep
MeSH Terms: interventions — cannabigerol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Cannabigerol (Experimental): 25 mg daily swallowable Cannabigerol tablets for 2 weeks, immediately followed by 50 mg daily swallowable Cannabigerol tablets for 2 weeks
  Interventions: Other: Cannabigerol
- Placebo (Placebo Comparator): 25 mg daily swallowable placebo tablets for 2 weeks, immediately followed by 50 mg daily swallowable placebo tablets for 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Cannabigerol — Cannabigerol is a non-psychoactive cannabinoid obtained from the cannabis plant.
  Arms: Active Cannabigerol
Other: Placebo — A placebo form of the same swallowable tablet with no cannabigerol
  Arms: Placebo

SUMMARY:
New methods for the treatment and support of Veterans experiencing sleep issues is critically needed. LEVEL's unique, targeted effects-based cannabis products provide a unique opportunity to study the therapeutic safety and efficacy of cannabigerol (a non-psychoactive cannabinoid) with a controlled dosage. Study participants will participate in an interventional, placebo-controlled, triple-blind pre-post study design. Participants will have a four-week run-in phase followed by an eight-week treatment phase with a CBG ProtabTM or placebo ProtabTM in a swallowable tablet form. During the study, participants will answer questions assessing their sleep, alcohol and drug use, and quality of life, among others. They will also wear a Fitbit Inspire 2 to collect biometric data.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* MOS Sleep Problems Index II > 30
* California resident
* Participants must own their own smartphone device to use for the study. Devices must meet the following criteria:
* Participants must be comfortable reading study instructions in English and communicating with study team in English
* Be willing to commit to study dosing, completing evaluation instruments, and following study protocol activities.
* If female and of childbearing potential, agree to use an effective form of birth control during study participation.

Exclusion Criteria:

* If using sleep medications, medication and dosage have not been changed in the past month and will remain unchanged for the duration of the study
* If using other psychotropic medications, medication and dosage have not been changed in the past 2 months, and will remain unchanged for the duration of the study
* Prior observation that the prospective participant has stopped breathing or observed choking/gasping during their sleep
* Previous diagnosis of sleep apnea (participant reported) without use of a CPAP (or similar PAP device) for at least the prior 4 weeks
* Currently in a Cognitive Behavioral Therapy for Insomnia (CBTI) program
* Women who are currently pregnant, trying to become pregnant, or breastfeeding
* Currently using CBG on a regular basis
* Participant has already participated in this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study (MOS) Sleep Problems Index II | 4 weeks
  Change in sleep quality from baseline scores as measured by the Medical Outcomes Study (MOS) Sleep Problems Index II after 4 weeks. Scores range from 0-100, with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
WHO-DAS-2.0-12 | 4 weeks
  Change in qualify of life from baseline scores on the World Health Organization Disability Assessment Schedule, Version 2.0 after 4 weeks. Scores range from 12-60, with higher scores indicating a worse outcome.

OTHER OUTCOMES:
Sleep Biometric Activity | 4 weeks
  Change in sleep Duration and quality from baseline to 4 weeks post-treatment, captured using a Fitbit Physical Activity Tracking Device
Activity Biometric Activity | 4 weeks
  Change in activity Duration and quality from baseline to 4 weeks post-treatment, captured using a Fitbit Physical Activity Tracking Device
Heart Rate Biometric Activity | 4 weeks
  Change in resting heart rate from baseline to 4 weeks post-treatment, captured using a Fitbit Physical Activity Tracking Device
Medical Outcomes Study (MOS) Sleep Problems Index II | 2 weeks
  Change in sleep quality from baseline scores as measured by the Medical Outcomes Study (MOS) Sleep Problems Index II after 2 weeks' treatment. Scores range from 0-100, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Virtual Site, Walnut, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Emerson CR, Webster CE, Daza EJ, Klamer BG, Tummalacherla M. Effect of Cannabigerol on Sleep and Quality of Life in Veterans: A Decentralized, Randomized, Placebo-Controlled Trial. Med Cannabis Cannabinoids. 2025 Dec 9;9(1):1-14. doi: 10.1159/000549902. eCollection 2026 Jan-Dec. PMID 41574318